CLINICAL TRIAL: NCT03208647
Title: Multi Center Case Control Study on Multiple Risk Factors of Aplastic Anemia Based on EDC Data Management Platform
Brief Title: Multi Center Case Control Study on Multiple Risk Factors of Aplastic Anemia
Acronym: MCSAA
Status: Completed | Type: Observational
Sponsor: Shengyun Lin (Other)
Responsible Party: Sponsor-Investigator, Shengyun Lin, chief, Zhejiang Provincial Hospital of TCM
Organization: Zhejiang Provincial Hospital of TCM (Other)
Other Study IDs: MCS-EDC-1802
Record Dates: First submitted 2016-07-18; First posted 2017-07-05 (Actual); Last update posted 2017-07-05 (Actual); Status verified 2017-07

CONDITIONS: Aplastic Anemia
Keywords: case-control study; Multiple risk factors
MeSH Terms: conditions — Anemia, Aplastic | interventions — Nuclear Receptor Subfamily 4, Group A, Member 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- AA Group: All the patients of AA group met a AA diagnostic criteria；
  Interventions: Other: AA or not
- Control Group: The control group were chosen from other departments who were under acute infection (such as pneumonia), acute abdominal emergency (such as appendicitis), cataract surgery;

INTERVENTIONS:
Other: AA or not — to study their risk factors
  Groups: AA Group

SUMMARY:
To ascertain the risk factors of AA in ZheJiang Province of China at the moment, especially the comprehensive multiple factors risks. The author conducted a case-control research included 338 AA cases and 1464 controls. Subjects were surveyed using same standard questionnaire including personal data, past histories of diseases, family history and histories of occupational and daily exposure to harmful substances. Single and multiple Logistic regression analyses were made using SPSS17.0 on the dates to study potential factors in the development of AA.

ELIGIBILITY:
Inclusion Criteria:

* All the patients of AA group met a AA diagnostic criteria；The control group were chosen from other departments who were under acute infection (such as pneumonia), acute abdominal emergency (such as appendicitis), cataract surgery;
* 1-65 years old, male or female;
* Sign the informed consent.

Exclusion Criteria:

* With myelodysplastic syndrome, leukaemia, multiple myeloma,megaloblastic anaemia, paroxysmal sleep hemoglobinuria disease blood disease, etc.
* History of tumor, radiation or chemotherapy, once accept the immunological therapy, autoimmune diseases or allergic disease patients;
* Patients with neurological diseases.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: All the patients of AA group met a AA diagnostic criteria；The control group were chosen from other departments who were under acute infection (such as pneumonia), acute abdominal emergency (such as appendicitis), cataract surgery; All cases had no history of tumor and radiation and chemotherapy, without receiving the immunological therapy; the control group cases without hematological diseases, autoimmune diseases, Fanconi anemia, congenital diseases, etc.
Sampling Method: Probability Sample
Enrollment: 1802 (Actual)
Dates: Start 2003-01-01; Primary Completion 2014-01-01 (Actual); Study Completion 2014-01-01 (Actual)

PRIMARY OUTCOMES:
the items about daily Exposures | January 2014
  Whether living or working near chemical factory or ionizing radiation, whether living in newly decorated apartments/house, having pets/livestock

SECONDARY OUTCOMES:
Individual Behaviours | January 2014
  Smoking (daily number of cigarettes )
Occupational Exposures | January 2014
  the duration of exposure to harmful substance(including industrial glue）
Individual Health Status | January 2014
  the time for the first onset of AA
Family disease history | January 2014
  Whether having the same disease, other blood diseases, malignant tumor

IPD SHARING:
Plan to Share IPD: No